CLINICAL TRIAL: NCT00003596
Title: A Phase III Randomized Study of 5-Fluorouracil, Mitomycin-C, and Radiotherapy Versus 5-Fluorouracil, Cisplatin, and Radiotherapy in Carcinoma of the Anal Canal
Brief Title: Chemotherapy Plus Radiation Therapy in Treating Patients With Stage II or Stage III Anal Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); Eastern Cooperative Oncology Group (Network); Cancer and Leukemia Group B (Network); SWOG Cancer Research Network (Network); North Central Cancer Treatment Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Treatment
Other Study IDs: RTOG-9811; CDR0000066667; CALGB-89808; ECOG-R9811; NCCTG-R9811; SWOG-R9811; GUMC-00125
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2017-01-04 (Estimated); Status verified 2016-12

CONDITIONS: Anal Cancer
Keywords: stage II anal cancer; stage III anal cancer; squamous cell carcinoma of the anus; cloacogenic carcinoma of the anus; basaloid carcinoma of the anus
MeSH Terms: conditions — Anus Neoplasms; Anal Canal Carcinoma | interventions — Cisplatin; Fluorouracil; Mitomycin; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: cisplatin
Drug: fluorouracil
Drug: mitomycin C
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug or combining radiation therapy with chemotherapy may kill more tumor cells. It is not yet known whether fluorouracil and mitomycin plus radiation therapy is more effective than fluorouracil and cisplatin plus radiation therapy for anal cancer.

PURPOSE: This randomized phase III trial is studying fluorouracil and mitomycin plus radiation therapy to see how well it works compared to fluorouracil and cisplatin plus radiation therapy in treating patients with stage II or stage III anal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the initial and total local and distant failure rates in patients with anal canal cancer treated with either fluorouracil (5-FU) plus mitomycin concurrently with radiotherapy or 5-FU plus cisplatin followed by 5-FU plus cisplatin concurrently with radiotherapy.
* Identify any differences in local control and colostomy rates at 2 years in patients treated with these regimens.
* Determine any difference in colostomy free, disease free, or overall survival in patients treated with these regimens.
* Compare the toxic effects of these regimens in these patients.
* Evaluate the prognostic effects of tumor markers P53 overexpression, human papilloma virus status, and enzyme HAP1 in patients treated with these regimens.

OUTLINE: This is a randomized study. Patients are stratified according to gender, nodal status (positive vs negative), and primary tumor size (greater than 2 cm to 5 cm vs greater than 5 cm). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive fluorouracil (5-FU) IV continuously over 96 hours beginning on days 1 and 29 and mitomycin IV on days 1 and 29 with concurrent radiotherapy.
* Arm II: Patients receive induction chemotherapy comprising 5-FU IV continuously over 96 hours beginning on days 1, 29, 57, and 85 and cisplatin IV over 1 hour on days 1, 29, 57, and 85. Beginning on day 57, patients receive concurrent radiotherapy.

In both arms, radiotherapy is administered daily, 5 days a week, for 5-6.5 weeks. Patients with T3, T4, or N+ lesions or T2 lesions with residual disease receive additional radiotherapy to a reduced field.

Patients are followed every 3 months for 1 year, every 6 months for 1 year, and then annually thereafter.

PROJECTED ACCRUAL: A total of 650 patients will be accrued for this study within 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed primary squamous, basaloid, or cloacogenic carcinoma of the anal canal, other than carcinoma in situ

  * T2-4, Any N, M0 (stage II or III)
* No local or regional recurrence after local excision or abdominal peritoneal resection

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 60-100%

Life expectancy:

* Not specified

Hematopoietic:

* WBC at least 4,000/mm^3
* Absolute neutrophil count at least 1,800/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 10 g/dL

Hepatic:

* Bilirubin less than 1.4 mg/dL

Renal:

* Creatinine no greater than 1.5 mg/dL OR
* Creatinine clearance at least 80 mL/min

Cardiovascular:

* No uncompensated heart disease
* No uncontrolled high blood pressure

Other:

* No AIDS
* No active systemic infection
* No uncontrolled diabetes
* No other prior malignancy within the past 5 years except nonmelanoma skin cancer
* No mental condition that would preclude study participation
* Not pregnant or nursing
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Prior epoetin alfa allowed in lieu of blood transfusions

Chemotherapy:

* At least 5 years since prior chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* At least 5 years since prior radiotherapy

Surgery:

* No prior surgery of anal canal except for biopsy of study site

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 682 (Actual)
Dates: Start 1998-10; Primary Completion 2005-10 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jaffer A. Ajani, MD, Study Chair — M.D. Anderson Cancer Center; Al B. Benson, MD, FACP, Study Chair — Robert H. Lurie Cancer Center; Joel E. Tepper, MD, Study Chair — UNC Lineberger Comprehensive Cancer Center; John S. MacDonald, MD, Study Chair — Beth Israel Comprehensive Cancer Center - West Side Campus; Michael G. Haddock, MD, Study Chair — Mayo Clinic
Locations (485):
- United States (484):
  - Comprehensive Cancer Center at University of Alabama at Birmingham, Birmingham, Alabama
  - Mobile Infirmary Medical Center, Mobile, Alabama
  - Alaska Regional Hospital, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Foundation for Cancer Research and Education, Phoenix, Arizona
  - CCOP - Mayo Clinic Scottsdale Oncology Program, Scottsdale, Arizona
  - Hembree Mercy Cancer Center at St. Edward Mercy Medical Center, Fort Smith, Arkansas
  - Alta Bates Comprehensive Cancer Center, Berkeley, California
  - Providence Saint Joseph Medical Center - Burbank, Burbank, California
  - Mills-Peninsula Health Services, Burlingame, California
  - Mount Diablo Regional Cancer Center, Concord, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - California Cancer Center - Woodward Park Office, Fresno, California
  - Marin Cancer Institute at Marin General Hospital, Greenbrae, California
  - Sutter Health Western Division Cancer Research Group, Greenbrae, California
  - Saint Rose Hospital, Hayward, California
  - Valley Memorial Hospital, Livermore, California
  - Loma Linda University Cancer Institute at Loma Linda University Medical Center, Loma Linda, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Providence Holy Cross Cancer Center, Mission Hills, California
  - Memorial Medical Center Cancer Services, Modesto, California
  - Leavey Cancer Center at Northridge Hospital Medical Center, Northridge, California
  - Highland General Hospital, Oakland, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Summit Medical Center, Oakland, California
  - Palo Alto Medical Foundation, Palo Alto, California
  - Pomona Valley Hospital Medical Center, Pomona, California
  - Radiological Associates of Sacramento Medical Group, Inc., Sacramento, California
  - University of California Davis Cancer Center, Sacramento, California
  - Naval Medical Center - San Diego, San Diego, California
  - California Pacific Medical Center - California Campus, San Francisco, California
  - J.C. Robinson, M.D. Regional Cancer Center, San Pablo, California
  - CCOP - Santa Rosa Memorial Hospital, Sana Rosa, California
  - Torrance Memorial Medical Center, Torrance, California
  - Sutter Solano Medical Center, Vallejo, California
  - Aurora Presbyterian Hospital, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Memorial Hospital Cancer Center, Colorado Springs, Colorado
  - Penrose Cancer Center at Penrose Hospital, Colorado Springs, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Presbyterian - St. Luke's Medical Center, Denver, Colorado
  - St. Joseph Hospital, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - CCOP - Colorado Cancer Research Program, Incorporated, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Front Range Cancer Specialists, Fort Collins, Colorado
  - St. Mary's Regional Cancer Center at St. Mary's Hospital and Medical Center, Grand Junction, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Hope Cancer Care Center at Longmont United Hospital, Longmont, Colorado
  - St. Mary-Corwin Regional Medical Center, Pueblo, Colorado
  - North Suburban Medical Center, Thorton, Colorado
  - Middlesex Hospital Cancer Center, Middletown, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - St. Francis Hospital, Wilmington, Delaware
  - Lombardi Cancer Center at Georgetown University Medical Center, Washington D.C., District of Columbia
  - Michael & Dianne Bienes Comprehensive Cancer Center at Holy Cross Hospital, Fort Lauderdale, Florida
  - 21st Century Oncology - Fort Myers, Fort Myers, Florida
  - Memorial Cancer Institute at Memorial Regional Hospital, Hollywood, Florida
  - Baptist Cancer Institute - Jacksonville, Jacksonville, Florida
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Ella Milbank Foshay Cancer Center at Jupiter Medical Center, Jupiter, Florida
  - University of Miami Sylvester Comprehensive Cancer Center, Miami, Florida
  - Baptist-South Miami Regional Cancer Program, Miami, Florida
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - Gulf Coast Cancer Treatment Center, Panama City, Florida
  - Tallahassee Memorial Hospital, Tallahassee, Florida
  - H. Lee Moffitt Cancer Center and Research Institute at University of South Florida, Tampa, Florida
  - Emory University Hospital - Atlanta, Altanta, Georgia
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Pearlman Comprehensive Cancer Center at South Georgia Medical Center, Valdosta, Georgia
  - Saint Alphonsus Cancer Care Center at Saint Alphonsus Regional Medical Center, Boise, Idaho
  - Mountain States Tumor Institute - Boise, Boise, Idaho
  - Saint Anthony's Hospital at Saint Anthony's Health Center, Alton, Illinois
  - Northwest Community Hospital, Arlington Heights, Illinois
  - Rush-Copley Cancer Care Center, Aurora, Illinois
  - Good Shepherd Hospital, Barrington, Illinois
  - St. Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital, Canton, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois
  - Creticos Cancer Center at Advocate Illinois Masonic Medical Center, Chicago, Illinois
  - Cancer Care Center at Advocate Good Samaritan Hospital, Downers Grove, Illinois
  - St. Anthony's Memorial Hospital, Effingham, Illinois
  - Eureka Hospital, Eureka, Illinois
  - Evanston Northwestern Health Care - Evanston Hospital, Evanston, Illinois
  - Galesburg Clinic, Galesburg, Illinois
  - Galesburg Cottage Hospital, Galesburg, Illinois
  - InterCommunity Cancer Center of Western Illinois, Galesburg, Illinois
  - Mason District Hospital, Havana, Illinois
  - Hinsdale Hematology Oncology Associates, Hinsdale, Illinois
  - Hopedale Medical Complex, Hopedale, Illinois
  - Joliet Oncology Hematology Associates, Limited - West, Joliet, Illinois
  - Kewanee Hospital, Kewanee, Illinois
  - McDonough District Hospital, Macomb, Illinois
  - Edward Hospital Cancer Center, Naperville, Illinois
  - BroMenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center, Normal, Illinois
  - Community Hospital of Ottawa, Ottawa, Illinois
  - Oncology Hematology Associates of Central Illinois - Ottawa, Ottawa, Illinois
  - Lutheran General Cancer Care Center, Park Ridge, Illinois
  - Cancer Treatment Center at Pekin Hospital, Pekin, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Proctor Hospital, Peoria, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Oncology/Hematology Associates of Central Illinois, P.C., Peoria, Illinois
  - OSF St. Francis Medical Center, Peoria, Illinois
  - Illinois Valley Community Hospital, Peru, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - Swedish American Hospital, Rockford, Illinois
  - St. Margaret's Hospital, Spring Valley, Illinois
  - Valley Cancer Center, Spring Valley, Illinois
  - Carle Cancer Center at Carle Foundation Hospital, Urbana, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - St. Francis Hospital and Health Centers, Beech Grove, Indiana
  - Bloomington Hospital, Bloomington, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Center for Cancer Therapy at LaPorte Hospital and Health Services, La Porte, Indiana
  - Saint Anthony Memorial Health Centers, Michigan City, Indiana
  - Cancer Center at Ball Memorial Hospital, Muncie, Indiana
  - Saint Joseph Regional Medical Center - Plymouth Campus, Plymouth, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Union Hospital, Terre Haute, Indiana
  - McFarland Clinic, P.C., Ames, Iowa
  - Saint Anthony Regional Hospital, Carroll, Iowa
  - St. Luke's Hospital, Cedar Rapids, Iowa
  - Cedar Rapids Oncology Associates, Cedar Rapids, Iowa
  - Mercy Cancer Center at Mercy Medical Center, Cedar Rapids, Iowa
  - Alegent Health Mercy Hospital, Council Bluffs, Iowa
  - Genesis Regional Cancer Center at Genesis Medical Center, Davenport, Iowa
  - Genesis Medical Center - West Campus, Davenport, Iowa
  - Mercy Capitol Hospital, Des Moines, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at John Stoddard Cancer Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at Mercy Cancer Center, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - Des Moines, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Lutheran Hospital, Des Moines, Iowa
  - Wendt Regional Cancer Center at Finley Hospital, Dubuque, Iowa
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - Mercy Cancer Center at Mercy Medical Center - North Iowa, Mason City, Iowa
  - Alegent Health Community Memorial Hospital, Missouri Valley, Iowa
  - Burgess Health Center, Onawa, Iowa
  - Siouxland Hematology-Oncology Associates, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Medical Oncology and Hematology Associates - West Des Moines, West Des Moines, Iowa
  - South Central Kansas Regional Medical Center, Arkansas City, Kansas
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, P.A. - El Dorado, El Dorado, Kansas
  - Kansas Masonic Cancer Research Institute at the University of Kansas Medical Center, Kansas City, Kansas
  - Cancer Center of Kansas - Kingman, Kingman, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Cancer Center of Kansas - Ottawa, Ottawa, Kansas
  - Cancer Center of Kansas, P.A. - Parsons, Parsons, Kansas
  - Pratt Cancer Center of Kansas, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates in Womens Health, Wichita, Kansas
  - Cancer Center of Kansas, P.A., Wichita, Kansas
  - Cancer Center of Kansas, P.A. - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Wesley Medical Center, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Cancer Treatment Center at the Medical Center - Bowling Green, Bowling Green, Kentucky
  - Central Baptist Hospital, Lexington, Kentucky
  - Markey Cancer Center at University of Kentucky Chandler Medical Center, Lexington, Kentucky
  - Merle M. Mahr Cancer Center at Regional Medical Center of Hopkins County, Madisonville, Kentucky
  - Louisiana State University Health Sciences Center - Monroe, Monroe, Louisiana
  - Tulane Cancer Center, New Orleans, Louisiana
  - Veterans Affairs Medical Center - Shreveport, Shreveport, Louisiana
  - Feist-Weiller Cancer Center at Louisiana State University Health Sciences, Shreveport, Louisiana
  - CancerCare of Maine at Eastern Maine Medial Center, Bangor, Maine
  - Central Maine Medical Center, Lewiston, Maine
  - Maine General Medical Center - Waterville, Waterville, Maine
  - DeCesaris Cancer Institute at Anne Arundel Medical Center, Annapolis, Maryland
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Union Hospital Cancer Center at Union Hospital, Elkton MD, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - Cancer Research Center at Boston Medical Center, Boston, Massachusetts
  - Bethke Cancer Center at Emerson Hospital, Concord, Massachusetts
  - Hudner Oncology Center at Saint Anne's Hospital, Fall River, Massachusetts
  - Cape Cod Hospital, Hyannis, Massachusetts
  - Newton - Wellesley Hospital, Newton, Massachusetts
  - South Suburban Oncology Center, Quincy, Massachusetts
  - Hickman Cancer Center at Bixby Medical Center, Adrian, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - St. Joseph Mercy Cancer Center at St. Joseph Mercy Hospital, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Battle Creek Health System, Battle Creek, Michigan
  - Mecosta County General Hospital, Big Rapids, Michigan
  - Josephine Ford Cancer Center at Henry Ford Health System, Detroit, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Great Lakes Cancer Institute at McLaren Regional Medical Center, Flint, Michigan
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - Lacks Cancer Center at Saint Mary's Mercy Medical Center, Grand Rapids, Michigan
  - Spectrum Health Cancer Care - Butterworth Campus, Grand Rapids, Michigan
  - Metropolitan Hospital, Grand Rapids, Michigan
  - Spectrum Health Hospital - Blodgett Campus, Grand Rapids, Michigan
  - Holland Community Hospital, Holland, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Borgess Medical Center, Kalamazooaa, Michigan
  - Upper Michigan Cancer Center at Marquette General Hospital, Marquette, Michigan
  - Hackley Hospital, Muskegon, Michigan
  - Northern Michigan Hospital, Petoskey, Michigan
  - Mercy Hospital, Port Huron, Michigan
  - Seton Cancer Institute - Saginaw, Saginaw, Michigan
  - Oncology Care Associates, P.L.L.C., Saint Joseph, Michigan
  - Providence Cancer Institute at Providence Hospital - Southfield Campus, Southfield, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - MeritCare Clinic - Bemidji, Bemidji, Minnesota
  - Brainerd Medical Center, Brainerd, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Cancer Care Center at St. Luke's Hospital, Duluth, Minnesota
  - CCOP - Duluth, Duluth, Minnesota
  - Miller-Dwan Medical Center, Duluth, Minnesota
  - St. Mary's - Duluth Clinic Cancer Center, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Mercy and Unity Cancer Center at Mercy and Unity Hospitals, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Meeker County Memorial Hospital, Litchfield, Minnesota
  - St. John's Hospital, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center - Minneapolis, Minneapolis, Minnesota
  - Fairview University Medical Center - University Campus, Minneapolis, Minnesota
  - Chippewa County - Montevideo Hospital, Montevideo, Minnesota
  - Hubert H. Humphrey Cancer Center at North Memorial Medical Center, Robbinsdale, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Adult and Pediatric Urology, P.L.L.P., Saint Cloud, Minnesota
  - CentraCare Clinic - River Campus, Saint Cloud, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Clinic, Saint Louis Park, Minnesota
  - Cancer Care Center at Regions Hospital, Saint Paul, Minnesota
  - St. Joseph's Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Cancer Center, Shakopee, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Woodwinds Hospital, Woodbury, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Veterans Affairs Medical Center - Jackson, Jackson, Mississippi
  - Regional Cancer Center at Singing River Hospital, Pascagoula, Mississippi
  - St. Francis Medical Center, Cape Girardeau, Missouri
  - Saint Luke's Hospital, Chesterfield, Missouri
  - Missouri Cancer Associates, Columbia, Missouri
  - Ellis Fischel Cancer Center at University of Missouri - Columbia, Columbia, Missouri
  - Southeast Missouri Regional Cancer Center at Southeast Missouri Hospital, Gape Girardeau, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - St. John's Regional Health Center, Springfield, Missouri
  - Hulston Cancer Center at Cox Medical Center South, Springfield, Missouri
  - Siteman Cancer Center at Barnes-Jewish Hospital, St Louis, Missouri
  - Missouri Baptist Cancer Center, St Louis, Missouri
  - CCOP - St. Louis-Cape Girardeau, St Louis, Missouri
  - Center for Cancer Care and Research, St Louis, Missouri
  - David C. Pratt Cancer Center at St. John's Mercy, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Sletten Regional Cancer Institute, Great Falls, Montana
  - Fremont Area Medical Center, Fremont, Nebraska
  - Cancer Center at the Good Samaritan Health Systems, Kearney, Nebraska
  - Bryan LGH Medical Center West, Lincoln, Nebraska
  - Cancer Resource Center - Lincoln, Lincoln, Nebraska
  - St. Elizabeth Regional Medical Center, Lincoln, Nebraska
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Methodist Hospital Cancer Center at Nebraska Methodist Hospital - Omaha, Omaha, Nebraska
  - Alegent Health - Immanuel Medical Center, Omaha, Nebraska
  - Bergan Mercy Medical Center, Omaha, Nebraska
  - Cancer Center at Creighton University Medical Center, Omaha, Nebraska
  - Midlands Cancer Center at Midlands Community Hospital, Papillion, Nebraska
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - Washoe Cancer Services at Washoe Medical Center - Reno, Reno, Nevada
  - Norris Cotton Cancer Center at Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Cancer Institute of New Jersey at the Cooper University Hospital, Camden, New Jersey
  - CCOP - Northern New Jersey, Hackensack, New Jersey
  - Monmouth Medical Center, Long Branch, New Jersey
  - South Jersey Healthcare Regional Cancer Center, Millville, New Jersey
  - Cancer Center at the Mountainside Hospital, Montclair, New Jersey
  - Fox Chase Virtua Health Cancer Program - Marlton, Mount Holly, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Atlantic City Medical Center - Mainland Division, Pomona, New Jersey
  - Booker Cancer Center at Riverview Medical Center, Red Bank, New Jersey
  - Community Medical Center, Toms River, New Jersey
  - Fox Chase Cancer Center at St. Francis Medical Center, Trenton, New Jersey
  - Capital Health System Regional Cancer Center, Trenton, New Jersey
  - Hematology-Oncology Associates, PC, Albuquerque, New Mexico
  - University of New Mexico Cancer Research and Treatment Center, Albuquerque, New Mexico
  - Lovelace Medical Center at Lovelace Sandia Health System, Albuquerque, New Mexico
  - SUNY Downstate Medical Center, Brooklyn, New York
  - New York Methodist Hospital, Brooklyn, New York
  - Finger Lakes Hematology and Oncology, Clifton Springs, New York
  - Louis Busch Hager Cancer Center at Mary Imogene Bassett Hospital, Cooperstown, New York
  - Catskill Regional Medical Center, Harris, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - New York Weill Cornell Cancer Center at Cornell University, New York, New York
  - Highland Hospital of Rochester, Rochester, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - CCOP - Syracuse Hematology-Oncology Associates of Central New York, P.C., Syracuse, New York
  - Crouse Hospital, Syracuse, New York
  - Veterans Affairs Medical Center - Syracuse, Syracuse, New York
  - Community General Hospital of Greater Syracuse, Syracuse, New York
  - Randolph Hospital, Asheboro, North Carolina
  - Blumenthal Cancer Center at Carolinas Medical Center, Charlotte, North Carolina
  - Presbyterian Cancer Center at Presbyterian Hospital, Charlotte, North Carolina
  - John Smith, Jr./Dalton McMichael Cancer Center at Morehead Memorial Hospital, Eden, North Carolina
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Wayne Radiation Oncology, Goldsboro, North Carolina
  - Moses Cone Regional Cancer Center at Wesley Long Community Hospital, Greensboro, North Carolina
  - Lenoir Memorial Cancer Center, Kinston, North Carolina
  - Annie Penn Cancer Center, Reidsville, North Carolina
  - Zimmer Cancer Center at New Hanover Regional Medical Center, Wilmington, North Carolina
  - Wilson Medical Center, Wilson, North Carolina
  - Forsyth Regional Cancer Center at Forsyth Medical Center, Winston-Salem, North Carolina
  - Bismarck Cancer Center, Bismarck, North Dakota
  - Medcenter One Health System, Bismarck, North Dakota
  - Mid Dakota Clinic, P.C., Bismarck, North Dakota
  - St. Alexius Medical Center, Bismarck, North Dakota
  - CCOP - MeritCare Hospital, Fargo, North Dakota
  - MeritCare Medical Group, Fargo, North Dakota
  - Altru Cancer Center at Altru Hospital, Grand Forks, North Dakota
  - Trinity Cancer Care Center, Minot, North Dakota
  - Akron City Hospital at Summa Health System, Akron, Ohio
  - McDowell Cancer Center at Akron General Medical Center, Akron, Ohio
  - University Hospitals Ireland Cancer Center at Mercy Medical Center, Canton, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Ireland Cancer Center at University Hospitals of Cleveland and Case Western Reserve University, Cleveland, Ohio
  - MetroHealth's Cancer Care Center at MetroHealth Medical Center, Cleveland, Ohio
  - Huron Hospital Cancer Care Center, Cleveland, Ohio
  - Euclid Hospital, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University, Columbus, Ohio
  - Riverside Methodist Hospital Cancer Care, Columbus, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Grant Riverside Cancer Services, Columbus, Ohio
  - Mount Carmel West Hospital, Columbus, Ohio
  - Doctors Hospital at Ohio Health, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Cancer Care Center, Dayton, Ohio
  - Veterans Affairs Medical Center - Dayton, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - St. Rita's Medical Center, Lima, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Strecker Cancer Center at Marietta Memorial Hospital, Marietta, Ohio
  - St. Luke's Hospital, Maumee, Ohio
  - Hillcrest Cancer Center at Hillcrest Hospital, Mayfield Heights, Ohio
  - Middletown Regional Hospital, Middletown, Ohio
  - Licking Memorial Cancer Care Program at Licking Memorial Hospital, Newark, Ohio
  - St. Charles Mercy Hospital, Oregon, Ohio
  - Cancer Research UK Medical Oncology Unit at Churchill Hospital & Weatherall Institute of Molecular Medicine - Oxford, Salem, Ohio
  - Firelands Regional Medical Center, Sandusky, Ohio
  - Mercy Medical Center Oncology Unit, Springfield, Ohio
  - Community Hospital of Springfield and Clark County, Springfield, Ohio
  - Promedica Cancer Center at Flower Hospital, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - Toledo Hospital, Toledo, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - Medical College of Ohio Cancer Institute, Toledo, Ohio
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - Toledo Clinic, Incorporated, Toledo, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - South Pointe Hospital Cancer Care Center, Warrensville Heights, Ohio
  - Mount Carmel Cancer Services at Mount Carmel St. Ann's Hospital, Westerville, Ohio
  - Cancer Treatment Center, Wooster, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - Genesis - Good Samaritan Hospital, Zanesville, Ohio
  - LaFortune Cancer Center at St. John Health System, Tulsa, Oklahoma
  - Natalie Warren Bryant Cancer Center at St. Francis Hospital, Tulsa, Oklahoma
  - Legacy Mount Hood Medical Center, Glesham, Oregon
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Comprehensive Cancer Center at Legacy Good Samaritan Hospital & Medical Center, Portland, Oregon
  - Providence Cancer Center at Providence Portland Medical Center, Portland, Oregon
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Institute of Oncology at Vilnius University, Portland, Oregon
  - Kaiser Permanente Health Care - Portland, Portland, Oregon
  - Cancer Institute at Oregon Health and Science University, Portland, Oregon
  - Salem Hospital Regional Cancer Center, Salem, Oregon
  - Legacy Meridian Park Hospital, Tualatin, Oregon
  - John and Dorothy Morgan Cancer Center at Lehigh Valley Hospital, Allentown, Pennsylvania
  - St. Luke's Hospital Cancer Center, Bethlehem, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Delaware County Regional Cancer Center at Delaware County Memorial Hospital, Drexel Hill, Pennsylvania
  - Penn State Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - St. Mary Regional Cancer Center, Langhorne, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - Cancer Center at Paoli Memorial Hospital, Paoli, Pennsylvania
  - Joan Karnell Cancer Center at Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Kimmel Cancer Center at Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Albert Einstein Cancer Center, Philadelphia, Pennsylvania
  - Allegheny Cancer Center at Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Mercy Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Western Pennsylvania Cancer Institute at Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - Pottstown Memorial Regional Cancer Center, Pottstown, Pennsylvania
  - St. Joseph Medical Center, Reading, Pennsylvania
  - Guthrie Medical Center - Sayre, Sayre, Pennsylvania
  - Mercy Hospital Cancer Center - Scranton, Scranton, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - Mount Nittany Medical Center, State College, Pennsylvania
  - Reading Hospital and Medical Center, West Reading, Pennsylvania
  - Geisinger Wyoming Valley Medical Center, Wilkes-Barre, Pennsylvania
  - CCOP - MainLine Health, Wynnewood, Pennsylvania
  - Lankenau Cancer Center at Lankenau Hospital, Wynnewood, Pennsylvania
  - Bon Secours St. Francis Health System, Greenville, South Carolina
  - Greenville Hospital System Cancer Center, Greenville, South Carolina
  - CCOP - Greenville, Greenville, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Sioux Valley Hospital and University of South Dakota Medical Center, Sioux Falls, South Dakota
  - Avera McKennan Hospital and University Health Center, Sioux Falls, South Dakota
  - Medical X-Ray Center, Sioux Falls, South Dakota
  - Baptist Centers for Cancer Care, Memphis, Tennessee
  - Harrington Cancer Center, Amarillo, Texas
  - St. Joseph Regional Cancer Center, Bryan, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - M.D. Anderson Cancer Center at University of Texas, Houston, Texas
  - Wilford Hall Medical Center, Lackland Air Force Base, Texas
  - Joe Arrington Cancer Research and Treatment Center, Lubbock, Texas
  - Veterans Affairs Medical Center - San Antonio (Murphy), San Antonio, Texas
  - Cancer Therapy and Research Center, San Antonio, Texas
  - University Hospital - San Antonio, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Cottonwood Hospital Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center - Provo, Provo, Utah
  - Utah Cancer Specialists at UCS Cancer Center, Salt Lake City, Utah
  - Huntsman Cancer Institute at University of Utah, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Dixie Regional Medical Center, St. George, Utah
  - Mountainview Medical, Berlin Corners, Vermont
  - Fletcher Allen Health Care - University Health Center Campus, Burlington, Vermont
  - Danville Regional Medical Center, Danville, Virginia
  - Virginia Oncology Associates - Hampton, Hampton, Virginia
  - Bon Secours Cancer Care at St. Mary's Hospital, Richmond, Virginia
  - St. Joseph Hospital Community Cancer Center, Bellingham, Washington
  - Olympic Hematology and Oncology, Bremerton, Washington
  - Providence Cancer Institute at Providence Everett Medical Center - Pacific Campus, Everett, Washington
  - Cancer Care Center at Skagit Valley Hospital, Mount Vernon, Washington
  - CCOP - Virginia Mason Research Center, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Group Health Central Hospital, Seattle, Washington
  - Harborview Medical Center, Seattle, Washington
  - Swedish Cancer Institute at Swedish Medical Center - First Hill Campus, Seattle, Washington
  - University Cancer Center at University of Washington Medical Center, Seattle, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Madigan Army Medical Center, Tacoma, Washington
  - Cancer Center at Southwest Washington Medical Center, Vancouver, Washington
  - Central Washington Hospital, Wenatchee, Washington
  - Wenatchee Valley Clinic, Wenatchee, Washington
  - Mary Babb Randolph Cancer Center at West Virginia University Hospitals, Morgantown, West Virginia
  - Camden-Clark Memorial Hospital, Parkersburg, West Virginia
  - Luther Mildelfort Hospital, Eau Claire, Wisconsin
  - Midelfort Clinic - Luther, Eau Claire, Wisconsin
  - Central Wisconsin Cancer Program at Agnesian Health Care, Fond du Lac, Wisconsin
  - Green Bay Oncology, Limited at St. Vincent Hospital, Green Bay, Wisconsin
  - St. Vincent Hospital, Green Bay, Wisconsin
  - Green Bay Oncology, Limited at St. Mary's Hospital, Green Bay, Wisconsin
  - St. Mary's Hospital Medical Center, Green Bay, Wisconsin
  - Gundersen Lutheran Cancer Center at Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
  - Bay Area Cancer Care Center at Bay Area Medical Center, Marinette, Wisconsin
  - Marshfield Clinic - Marshfield Center, Marshfield, Wisconsin
  - Community Memorial Hospital, Menomonee Falls, Wisconsin
  - Vince Lombardi Cancer Clinic at St. Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin Cancer Center, Milwaukee, Wisconsin
  - Veterans Affairs Medical Center - Milwaukee (Zablocki), Milwaukee, Wisconsin
  - All Saints Cancer Center at All Saints Healthcare, Racine, Wisconsin
  - West Allis Memorial Hospital, West Allis, Wisconsin
- Pretoria Academic Hospital, Pretoria, South Africa

REFERENCES:
- [Background] Ben-Josef E, Moughan J, Ajani JA, Flam M, Gunderson L, Pollock J, Myerson R, Anne R, Rosenthal SA, Willett C. Impact of overall treatment time on survival and local control in patients with anal cancer: a pooled data analysis of Radiation Therapy Oncology Group trials 87-04 and 98-11. J Clin Oncol. 2010 Dec 1;28(34):5061-6. doi: 10.1200/JCO.2010.29.1351. Epub 2010 Oct 18. PMID 20956625
- [Background] Glynne-Jones R, Mawdsley S. Anal cancer: is neoadjuvant cisplatin chemotherapy or chemoradiotherapy friend or foe? Nat Clin Pract Oncol. 2008 Dec;5(12):692-3. doi: 10.1038/ncponc1258. Epub 2008 Oct 14. PMID 18852720
- [Result] Gunderson LL, Winter KA, Ajani JA, et al.: Long-term update of U.S. GI intergroup RTOG 98-11 phase III trial for anal carcinoma: disease-free and overall survival with RT+5FU-mitomycin versus RT+5FU-cisplatin. [Abstract] J Clin Oncol 29 (Suppl 15): A-4005, 2011.
- [Result] Ajani JA, Winter KA, Gunderson LL, Pedersen J, Benson AB 3rd, Thomas CR Jr, Mayer RJ, Haddock MG, Rich TA, Willett CG. Prognostic factors derived from a prospective database dictate clinical biology of anal cancer: the intergroup trial (RTOG 98-11). Cancer. 2010 Sep 1;116(17):4007-13. doi: 10.1002/cncr.25188. PMID 20564111
- [Result] Gunderson LL, Moughan J, Ajani JA, et al.: Anal carcinoma: Impact of TN category of disease on survival, disease relapse, and colostomy failure in U.S. GI Intergroup RTOG 98-11 phase III trial. [Abstract] American Society of Clinical Oncology 2010 Gastrointestinal Cancers Symposium, 22-24 January 2010, Orlando, Florida. A-285, 2010.
- [Result] Ajani JA, Winter KA, Gunderson LL, Pedersen J, Benson AB 3rd, Thomas CR Jr, Mayer RJ, Haddock MG, Rich TA, Willett CG. US intergroup anal carcinoma trial: tumor diameter predicts for colostomy. J Clin Oncol. 2009 Mar 1;27(7):1116-21. doi: 10.1200/JCO.2008.19.6857. Epub 2009 Jan 12. PMID 19139424
- [Result] Ajani JA, Winter KA, Gunderson LL, Pedersen J, Benson AB 3rd, Thomas CR Jr, Mayer RJ, Haddock MG, Rich TA, Willett C. Fluorouracil, mitomycin, and radiotherapy vs fluorouracil, cisplatin, and radiotherapy for carcinoma of the anal canal: a randomized controlled trial. JAMA. 2008 Apr 23;299(16):1914-21. doi: 10.1001/jama.299.16.1914. PMID 18430910
- [Result] Ajani JA, Winter KA, Gunderson LL, et al.: Intergroup RTOG 98-11: a phase III randomized study of 5-fluorouracil (5-FU), mitomycin, and radiotherapy versus 5-fluorouracil, cisplatin and radiotherapy in carcinoma of the anal canal. [Abstract] J Clin Oncol 24 (Suppl 18): A-4009, 2006.
- [Result] Gunderson LL, Winter KA, Ajani JA, et al.: Intergroup RTOG 9811 phase III comparison of chemoradiation with 5-FU and mitomycin vs 5-FU and cisplatin for anal canal carcinoma: impact on disease-free, overall and colostomy-free survival. [Abstract] Int J Radiat Oncol Biol Phys 66 (3 Suppl 1): A-43, S24, 2006.
- [Derived] Gunderson LL, Winter KA, Ajani JA, Pedersen JE, Moughan J, Benson AB 3rd, Thomas CR Jr, Mayer RJ, Haddock MG, Rich TA, Willett CG. Long-term update of US GI intergroup RTOG 98-11 phase III trial for anal carcinoma: survival, relapse, and colostomy failure with concurrent chemoradiation involving fluorouracil/mitomycin versus fluorouracil/cisplatin. J Clin Oncol. 2012 Dec 10;30(35):4344-51. doi: 10.1200/JCO.2012.43.8085. Epub 2012 Nov 13. PMID 23150707